CLINICAL TRIAL: NCT06073808
Title: The Role of Amnion Membrane Allografts in Nipple Preservation After Nipple Sparing Mastectomy: A Double-Blinded Randomized Controlled Trial
Brief Title: The Role of Amnion Membrane Allografts in Nipple Preservation
Acronym: AmnioFix
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Dung Nguyen, Clinical Professor, Director of Breast Reconstruction, Director of Adult Plastics and Reconstructive Clinic, Associate Director of Microsurgery, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 71564
Record Dates: First submitted 2023-09-09; First posted 2023-10-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Mastectomy; Gender Affirmation Surgery; Nipple Sparing Mastectomy; Prophylactic Mastectomy; Benign Breast Condition
Keywords: nipple sparing mastectomy; gender affirming surgery

STUDY DESIGN:
Intervention Model Description: Each patient will serve as their own control: one breast will receive the control device, and the other will receive the study device.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Assess dHACM viability (Experimental): Implantation of dHACM in patients during Nipple Sparing Mastectomy; test arm. The device will be implanted in one breast per patient during bilateral nipple sparing mastectomy.
  Interventions: Device: AmnioFix dehydrated Human Amnion/Chorion Membrane Allograft
- Assess dHACM effectiveness against control device (Active Comparator): Implantation of control device in patients during Nipple Sparing Mastectomy; control arm. The device will be implanted in one breast per patient during bilateral nipple sparing mastectomy.
  Interventions: Device: Control Device

INTERVENTIONS:
Device: AmnioFix dehydrated Human Amnion/Chorion Membrane Allograft — Dehydrated human amnion/chorion membrane (dHACMs) allografts have recently been identified as an easy-to-use treatment alternative for management of chronic wounds. These commercially available allografts contain concentrated cytokines and growth factors known to promote wound healing. Preclinical studies suggest that dHACM allografts provide a complex, biologically-driven mechanism to promote soft tissue repair and regeneration, including stimulation of mesenchymal stem cell migration and dermal fibroblast proliferation, establishment of a supportive inflammatory environment, and restoration of extracellular matrix integrity with positive tissue architecture remodeling. Clinically, dHACM allografts have been shown to improve healing time and wound closure rates in chronic wound patients. However, no study to date has evaluated the impact of dHACM allografts on nipple necrosis following NSM.
  Other Names: AmnioFix
  Arms: Assess dHACM viability
Device: Control Device — Control device will be applied to non-experimental breast. Each patient will serve as their own control.
  Arms: Assess dHACM effectiveness against control device

SUMMARY:
The overall objective of this proposal is to conduct a randomized-controlled study to determine whether treatment with dehydrated human amnion/chorion membrane (dHACMs) allografts can improve NAC viability in patients undergoing nipple sparing mastectomy (NSM). dHACM allografts are commercially available tissue membranes with biocompatible extracellular matrix and growth factors that have been shown to improve wound healing in patients with chronic and lower extremity wounds. To date, no study has evaluated the impact of dHACMs on NAC preservation following NSM. Investigators hypothesize that subareolar surgical implantation of dHACM allografts at time of NSM will reduce NAC necrosis and improve viability.

DETAILED DESCRIPTION:
This proposal will be the first clinical trial to evaluate the clinical efficacy of dHACM allografts in NSM. The topic of study not only addresses a critically unmet need in the field of plastic surgery, but also maintains exceptional scientific and clinical merit. This study would be the first to establish dHACM allografts as a novel, innovative, and biologically-based adjunctive mechanism to improve vascularity and wound healing following NSM. Such findings would not only provide the evidence-base for widespread implementation of dHACM allografts in the surgical management of breast patients, but also serve as a catalyst to study the clinical efficacy of these allografts in other plastic surgical patient cohorts. Overall, this proposal aims to serve as a successful translational model incorporating scalable, biologically-based regenerative therapies in a surgical population.

Nipple necrosis is a major complication after nipple sparing mastectomy, a procedure that is commonly performed in the human population for gender reassignment surgery and for breast cancer prevention. This study will assess the efficacy of dHACMs can improve nipple viability after NSM.

ELIGIBILITY:
Inclusion Criteria:

* Biologically female with documented diagnosis of gender dysphoria, desire to undergo gender affirming surgery (female-to-male) NSM, and age 15 years of age or older.
* Biological female, age 18 to 75 years old, who desire to undergo bilateral prophylactic NSM for nonmalignant breast conditions or to reduce the risk of breast cancer.

Exclusion Criteria:

* Current steroid use
* Known connective tissue disorder
* Known neuropathy
* Known history of breast cancer
* History of breast radiotherapy
* Pregnant or nursing

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Nipple Necrosis in patients who receive dHACM during nipple sparing mastectomy (NSM) | through study completion, an average of 3 months post op
  The primary endpoint of this study is number of nipples with necrosis as defined by dark blue or black nipple discoloration, ultimately resulting in scabs or open wounds up to 3 months post-operatively.

SECONDARY OUTCOMES:
Rate of Nipple Healing | through study completion, an average of 3 months post op
  Number of nipples that have healed per clinician assessment.
Degree of nipple loss | through study completion, an average of 3 months post op
  Number of nipples partially or wholly lost to necrosis.
Nipple perfusion | through study completion, an average of 3 months post op
  Perfusion of blood in the nipple assessed via indocyanine green (ICG)-SPY technology.
Aesthetic satisfaction scale score; scale used is a likert scale (very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, very dissatisfied | through study completion, an average of 3 months post op
  Participant-rated satisfaction.
Number of Participants with Nipple Sensation | through study completion, an average of 3 months post op
  Participants indicated whether they have nipple sensation (innervation) (Y/N).

CONTACTS AND LOCATIONS:
Overall Officials: Dung Nguyen, MD, PharmD, Principal Investigator — Stanford University
Locations (1):
- Division of Plastic & Reconstructive Surgery, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No